CLINICAL TRIAL: NCT01321242
Title: Observational Non-interventional Study - Epidemiological Survey "AchievemenT of Goal Resting HEart Rate on Beta-blockers in Patients With Stable angiNA and Hypertension in Routine Practice"
Brief Title: Achievement of Goal Resting Heart Rate on B-blockers in Patients With Stable Angina and Hypertension
Acronym: Athena
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CRU-ATC-2011/1
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Stable Angina; Hypertension
Keywords: Resting heart rate; Stable Angina; Hypertension; beta-blockers
MeSH Terms: conditions — Angina, Stable; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- achieving resting HR goals: Patient population will be comprised of typical for cardiological practice sample of patients with Coronary Heart Disease and arterial hypertension administered beta-blockers, subjects achieving resting HR goals, according to ACC/AHA/ACP-ASIM Guidelines
- non-achieving HR goals: Patient population will be comprised of typical for cardiological practice sample of patients with Coronary Heart Disease and arterial hypertension administered beta-blockers, subjects non-achieving HR goals, according to ACC/AHA/ACP-ASIM Guidelines

SUMMARY:
This is a multicenter survey of Russian data on target heart rate achievement in patients with stable angina and arterial hypertension who are currently treated with beta-blockers for at least 2 months and with no dose change for a minimum of 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Stable angina I-III class by the Canadian Cardiovascular Society Classification and concomitant primary hypertension
* Subject is on beta-blockers treatment for at least 2 months prior to inclusion into survey, with no dose change for a minimum of 4 weeks

Exclusion Criteria:

* Use of phenylalkylamine and benzothiazepine calcium channel blockers
* Hemodynamic significant mitral and aortic valve disease
* Acute myocardial infarction and unstable angina within 3 months before enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Establish the proportion of patients with stable angina and hypertension on beta-blockers reaching the resting HR goals according to ACC/AHA/ACP-ASIM* Guidelines | 1 visit within 5 month
  *American College of Cardiology (ACC)/American Heart Association (AHA)/American College of Physicians (ACP-ASIM)

SECONDARY OUTCOMES:
Establish the mean dose of each beta-blocker in patients who achieved and not achieved resting HR goals | 1 visit within 5 month
Compare quality of life in patients who achieved and non achieved resting HR goals | 1 visit within 5 month
To estimate the correlation between achievement of resting HR goals according to ACC/AHA/ACP-ASIM Guidelines for the management of patients | 1 visits within 5 month

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Stepanov, Study Director — AstraZeneca; Z.D. Kobalava, Principal Investigator — The Russian Peoples' Friendship University, Municipal Clinical Hospital #64
Locations (6):
- Russia (6):
  - Research Site, Moscow
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Ulyanovsk
  - Research Site, Yekaterinburg

REFERENCES:
- [Derived] Kobalava Z, Khomitskaya Y, Kiyakbaev G; ATHENA trial investigators. AchievemenT of target resting HEart rate on beta-blockers in patients with stable angiNA and hypertension (ATHENA) in routine clinical practice in Russia. Curr Med Res Opin. 2014 May;30(5):805-11. doi: 10.1185/03007995.2013.874993. Epub 2014 Jan 17. PMID 24400847